CLINICAL TRIAL: NCT06316180
Title: The Use of Drospirenone/Estetrol in Random Start Rapid Preparation of Endometrium Before Office Hysteroscopic Polypectomies: a Multicenter, Prospective, Randomized Study
Brief Title: The Use of Drospirenone/Estetrol in Random Start Rapid Endometrial Preparation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Palermo (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea Etrusco, Principal investigator, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DROVPREP
Record Dates: First submitted 2024-03-07; First posted 2024-03-18 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Endometrial Polyp; Endometrial Diseases
Keywords: Hysteroscopy; Endometrial Preparation
MeSH Terms: conditions — Uterine Diseases | interventions — drospirenone; Estetrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Patients with endometrial polyps undergone hysteroscopic polipectomy without endometrial preparation.
- Intervention (Active Comparator): Patients with endometrial polyps underwent hysteroscopic polipectomy after starting 14-day treatment with oral drospirenone/estetrol 3mg/14.2mg at any time of the menstrual cycle.
  Interventions: Drug: drospirenone/estetrol 3mg/14.2mg

INTERVENTIONS:
Drug: drospirenone/estetrol 3mg/14.2mg — Hysteroscopic polipectomy after starting 14-day treatment with oral drospirenone/estetrol 3mg/14.2mg at any time of the menstrual cycle.
  Arms: Intervention

SUMMARY:
The presence of a thin endometrium plays an important role in enabling the best conditions for hysteroscopic surgery. Recently, for this purpose, many studies have evaluated the effect of preoperative administration of a variety of drugs. We explored the efficacy of random started 14-day administration of drospirenone/estetrol, in rapid preparation of endometrium for hysteroscopic polypectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with endometrial polyps.

Exclusion Criteria:

* Patients with other endometrial pathologies.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Quality of endometrial preparation | Intraoperatively
  Quality of endometrial preparation assessed visually intraoperatively by the surgeon using a visual analog scale from 0 to 5.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Andrea Etrusco, Palermo
  - Marco Monti, Rome